CLINICAL TRIAL: NCT00911573
Title: A Phase 3, Multicenter, Randomized, Double-Blind Study To Evaluate The Safety And Efficacy Of Tigecycline Versus Comparator (Clindamycin Or Vancomycin) For The Treatment Of Complicated Skin And Skin Structure Infections, Including Those Due To MRSA, In Pediatric Subject Ages 8 To 17 Years Old
Brief Title: Study Evaluating Tigecycline Versus Clindamycin Or Vancomycin On Complicated Skin And Skin Structure Infections Including Those Due To Methicillin-Resistant Staphylococcus Aureus (MRSA) In Pediatric Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3074K4-3339; B1811002
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Skin Diseases; Infection
Keywords: pediatry; children; skin; bacteria; MRSA
MeSH Terms: conditions — Skin Diseases; Infections | interventions — Tigecycline; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Tigecycline
  Interventions: Drug: Tigecycline
- B (Active Comparator): Clindamycin (or Vancomycin if needed)
  Interventions: Drug: Clindamycin (or Vancomycin if needed)

INTERVENTIONS:
Drug: Tigecycline — 50 mg IV every 12 hours up to 14 days
  Other Names: Tygacil
  Arms: A
Drug: Clindamycin (or Vancomycin if needed) — For clindamycin 10mg/kg (not to exceed 900mg) IV every 8 hours up to 14 days. For vancomycin 15mg/kg (not to exceed 2g/day and adjusted as needed for renal impairment) IV every 8 hours
  Arms: B

SUMMARY:
The main purpose of this study is to compare the safety and efficacy of tigecycline versus clindamycin (including subjects treated with vancomycin) in pediatric subjects (aged 8 to 17 years) with complicated skin and skin structure infections (cSSSI), including those caused by methicillin-resistant staphylococcus aureus (MRSA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 8 to 17 years old. Children with bone maturation less than 8 years old should be enrolled with caution due to potential risk of tooth discoloration.
* Have a diagnosis of a serious infection requiring hospitalization and administration of IV antibiotic therapy.
* complicated skin and skin structure infections (cSSSI) requiring significant surgical intervention or involving deeper soft tissue with the presence of at least one sign of systemic infection

Exclusion Criteria:

* Subject with any concomitant illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and/or completion of the study, or could preclude the evaluation of the subject's response (e.g., life expectancy < 30 days).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate at the test-of-cure visit for the 2 co-primary populations: clinically evaluable and clinically modified intent to treat populations | 15-37 days

SECONDARY OUTCOMES:
Microbiologic response at the subject level and at the pathogen level measured at intravenous last day of therapy (IV LDOT), test-of-cure (TOC) and follow-up (FUP) visits | 5-49 days
Clinical cure rates by baseline pathogen (including MRSA) at test-of-cure (TOC) visit | 15-37 days
Clinical response and microbiological response at the subject level for subjects with monomicrobial and polymicrobial infections at test-of-cure (TOC) visit | 15-37 days
Development of decreased susceptibility | 5-50 days
Clinical response and microbial response at subject level by baseline pathogen and minimum inhibitory concentration (MIC) values at test-of-cure (TOC) visit | 15-37 days
Susceptibility data by pathogen | 5-50 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074K4-3339&StudyName=Study%20Evaluating%20Tigecycline%20Versus%20Clindamycin%20Or%20Vancomycin%20On%20Complicated%20Skin%20And%20Skin%20Structure%20Infections%20Including%20Those%20Due%20To%20